CLINICAL TRIAL: NCT06153290
Title: Blinding Integrity Following a Single Session of Simulated or Genuine High Velocity, Low Amplitude (HVLA) Manual Chiropractic Adjustments: a Randomized Controlled Proof-of-concept Trial
Brief Title: Patient Perceptions Following a Single Session of Simulated or Genuine HVLA Manual Chiropractic Adjustments
Acronym: SHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Life University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: I-0026
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Subluxation
Keywords: randomized; sham-controlled; chiropractic; blinding
MeSH Terms: conditions — Joint Dislocations | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Intervention Model Description: Randomized, sham-controlled, proof-of-concept trial
Who Masked: Participant
Masking Description: Single-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genuine/real (Experimental): 15 participants receiving genuine/real chiropractic adjustment
  Interventions: Procedure: Chiropractic adjustment
- Simulated/sham (Sham Comparator): 15 participants receiving simulated/sham "adjustment"
  Interventions: Procedure: Sham adjustment

INTERVENTIONS:
Procedure: Chiropractic adjustment — A single-session of genuine/real high-velocity, low-amplitude (HVLA) manual chiropractic adjustments to various regions of the spine (i.e., cervical, thoracic, lumbo-pelvic)
  Arms: Genuine/real
Procedure: Sham adjustment — A single-session of simulated/sham high-velocity, low-amplitude (HVLA) manual chiropractic adjustments to various regions of the spine (i.e., cervical, thoracic, lumbo-pelvic)
  Arms: Simulated/sham

SUMMARY:
The primary aim of this trial is to assess blinding following simulated/sham or genuine/real high velocity, low amplitude (HVLA) manual chiropractic adjustments.

DETAILED DESCRIPTION:
The primary aim of this trial is to assess blinding following simulated/sham or genuine/real high velocity, low amplitude (HVLA) manual chiropractic adjustments. Briefly, 30 eligible participants will be randomized (1:1 ratio) to receive a single session of either simulated/sham or genuine/real chiropractic spinal adjustments and be given a brief survey immediately following their session and 48 hours later that captures their perceptions and experiences regarding the intervention they received. This study is intended to inform a future multi-session, randomized, sham-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age

Exclusion Criteria:

* History of stroke or transient ischemic attack or current symptoms including dizziness or vertigo, tinnitus (ringing in the ears), or visual, sensory, or motor disturbances
* New pattern headache complaint
* Recent whiplash injury (within 12 months)
* Cervical fracture/dislocation
* Disc problem with radiating symptoms to the arms or legs
* Severe degenerative joint disease in the spine
* Connective tissue disorder
* Primary fibromyalgia
* Metabolic or metaplastic bone disease
* History of cervical, thoracic, or lumbar spine surgery
* Uncontrolled high blood pressure or vascular disease
* Current use of anticoagulant therapy
* Doctor of Chiropractic (DC) or a DC student in 5th quarter or above
* Present, self-reported pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Participant blinding | Immediately after intervention
  The blinding index is scaled to an internal of -1 to +1, +1 being complete lack of blinding, 0 being consistent with perfect blinding, -1 indicating opposite guessing which may be related to unblinding.
Participant blinding | 48 hours after intervention
  The blinding index is scaled to an internal of -1 to +1, +1 being complete lack of blinding, 0 being consistent with perfect blinding, -1 indicating opposite guessing which may be related to unblinding.

CONTACTS AND LOCATIONS:
Overall Officials: Tyson Perez, DC, PhD, Principal Investigator — Life University
Locations (1):
- Dr. Sid E. Williams Center for Chiropractic Research, Marietta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/90/NCT06153290/ICF_000.pdf